CLINICAL TRIAL: NCT04495894
Title: A Pilot Study of Biomarker Evaluation and Safety of Pre-Incisional Ketorolac for Patients Undergoing Surgical Resection for Non-Small Cell Lung Cancer and Renal Cell Carcinoma
Brief Title: Pre-Incisional Ketorolac for Patients Undergoing Surgery for Non-Small Cell Lung Cancer and Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated after interim analyses showed no benefits.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Viraj Master, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00000205
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer; Renal Cell Carcinoma
Keywords: Surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell | interventions — Ketorolac Tromethamine; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Preoperative Ketorolac For Participants with Non-small Cell Lung Carcinoma (NSCLC) (Experimental): Participants randomized to receive ketorolac prior to surgery for stage I/II non-small cell lung carcinoma (NSCLC). Participants receive standard-of-care surgery. Open, video-assisted thoracic surgery, laparoscopy, or robotic surgery are allowed. Standard anesthesia is administered.
  Interventions: Drug: Preoperative Ketorolac
- Control Group For Participants with Non-small Cell Lung Carcinoma (NSCLC) (No Intervention): Participants randomized to the control group receiving the standard of care during surgery for stage I/II non-small cell lung carcinoma (NSCLC). Open, video-assisted thoracic surgery, laparoscopy, or robotic surgery are allowed. Standard anesthesia is administered. The concurrent control group is to obtain untreated biologic samples for biologic correlative studies and secondary endpoints.
- Preoperative Ketorolac For Participants with renal cell carcinoma (RCC) (Experimental): Participants randomized to receive ketorolac prior to surgery for stage III renal cell carcinoma (RCC). Participants receive standard-of-care surgery. Open, video-assisted thoracic surgery, laparoscopy, or robotic surgery are allowed. Standard anesthesia is administered.
  Interventions: Drug: Preoperative Ketorolac
- Control Group For Participants with renal cell carcinoma (RCC) (No Intervention): Participants randomized to the control group receiving the standard of care during surgery for stage III renal cell carcinoma (RCC). Open, video-assisted thoracic surgery, laparoscopy, or robotic surgery are allowed. Standard anesthesia is administered. The concurrent control group is to obtain untreated biologic samples for biologic correlative studies and secondary endpoints.

INTERVENTIONS:
Drug: Preoperative Ketorolac — 30 mg ketorolac will be administered intravenously 30 minutes prior to incision.
  Other Names: Acular; Acuvail
  Arms: Preoperative Ketorolac For Participants with Non-small Cell Lung Carcinoma (NSCLC); Preoperative Ketorolac For Participants with renal cell carcinoma (RCC)

SUMMARY:
This is a pilot study of biomarker evaluation and safety of pre-incisional ketorolac for patients undergoing surgical resection for non-small cell lung cancer and renal cell carcinoma. There is significant promise in the use of preoperative ketorolac to decrease the inflammatory response after surgical resection of tumors, thereby potentially reducing the risk of distant metastatic tumor spread and improving survival. This research will advance scientific knowledge by studying the safety of a preoperative dose of ketorolac prior to major surgical resection, which needs to be assessed prior to proceeding with a larger phase II study designed to evaluate traditional efficacy endpoints such as recurrence and overall survival.

DETAILED DESCRIPTION:
Surgical resection is a cornerstone of standard-of-care treatment for early-stage non-small cell lung carcinoma (NSCLC) and renal cell carcinoma (RCC). Yet despite optimal treatment, many of these patients will develop cancer recurrence within the first few years. For example, the 5-year survival rate for patients with stage I/II NSCLC is only around 55%. As a result, more effective treatments that decrease cancer recurrence and increase survival are still needed.

Surgery induces inflammation, immunosuppression and angiogenesis. Although these processes are important for wound healing in response to tissue injury caused by surgery, they also support the survival, growth and dissemination of any remaining cancer cells and can lead to systemic recurrence soon after surgery. Surgical trauma increases the production of prostaglandins and thromboxanes, which have tumor-promoting and immunosuppressive activities, and reduces the activity of natural killer cells, which impairs the ability of the immune system to keep cancer cells in check. However, if given just before tissue injury, non-steroidal anti-inflammatory drugs (NSAIDs) may be able to block the production of prostaglandins/thromboxanes and boost the activity of natural killer cells, and thereby decrease the risk of cancer recurrence. NSAIDs such as ketorolac are already routinely given to cancer patients postoperatively for pain management and are sometimes given intraoperatively (immediately before or during surgery) to prevent postoperative pain. A retrospective clinical analysis found that intraoperative intravenous ketorolac or diclofenac (another NSAID), when added to standard of care for patients with stage I/II NSCLC, was associated with decreased risks of distant recurrence and mortality.

In this study, patients with NSCLC or RCC will be screened and recruited during the preoperative period by the responsible medical and surgical team. Participants will be randomized on the day of surgery to either the preoperative ketorolac group or a concurrent control group who will not receive preincisional ketorolac. Participants will be followed for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Pathology-proven or suspected stage 1 or 2 NSCLC and Stage 3 tumor stage 3, node stage 0 (T3N0) RCC, that require surgical resection as the treatment of choice
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Ability to understand and the willingness to sign an informed written consent

Exclusion Criteria:

* Individuals with pure lung ground-glass opacity (GGO) lesions or mixed GGO with <50% solid component
* Patients undergoing pneumonectomy
* History of cancer in the 3 years prior to surgery (except for basal-cell carcinoma of the skin or cervical neoplasia).
* Contraindication for NSAIDs, including peptic ulcer disease, preoperative chronic kidney disease with estimated glomerular filtration rate (eGFR) <45, allergies or intolerance to NSAIDs, coagulation disorder, or age > 80 years
* Having taken an NSAID within 5 days prior to surgery
* Immunocompromised status
* Refusal or inability to understand the protocol and consent form or to receive follow-up in line with the recommendations
* Preoperative hemoglobin < 9.0

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viraj Master, MD, PhD, Principal Investigator — Emory University; Onkar Khullar, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Clinic, Emory University Hospital Midtown, Emory University Hospital, and the Winship Cancer Institute in Atlanta, Georgia, USA. Participant enrollment began August 24, 2020 the final study assessment occurred February 1, 2024.
Period: Overall Study
Arm/Group | Preoperative Ketorolac For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Control Group For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Preoperative Ketorolac For Participants With Renal Cell Carcinoma (RCC) | Control Group For Participants With Renal Cell Carcinoma (RCC)
Started (Participants who passed screening and were randomized to a study arm) | 16 | 6 | 33 | 13
Participants Who Started the Study Activities of Ketorolac Administration (if Assigned) and Surgery | 14 | 6 | 28 | 10
Completed | 14 | 6 | 28 | 10
Not Completed | 2 | 0 | 5 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 3
Not completed — Early termination | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes participants who started the study activities of administration of ketorolac (for participants in a ketorolac study arm) and had their standard of care surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative Ketorolac For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Control Group For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Preoperative Ketorolac For Participants With Renal Cell Carcinoma (RCC) | Control Group For Participants With Renal Cell Carcinoma (RCC) | Total
Number analyzed (Participants) | 14 | 6 | 28 | 10 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (6.2) | 61.2 (8.9) | 59.9 (13.9) | 62.2 (13.6) | 62.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 10 | 2 | 26
  Male | 5 | 1 | 18 | 8 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 6 | 17 | 8 | 45
  Unknown or Not Reported | 0 | 0 | 10 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 4 | 3 | 10
  White | 12 | 4 | 17 | 6 | 39
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 6 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 6 | 28 | 10 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving a Blood Transfusion
Description: Hemorrhagic side effects among participants receiving ketorolac preoperatively will be assessed as the need for blood transfusions before being discharged from the hospital after surgery. The need for a blood transfusion is defined as needing two or more units of blood, which are not related to vascular injury due to technical considerations or complications, as determined by the operating surgeon.
Time Frame: Prior to Hospital Discharge (up to 13 days post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Ketorolac For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Control Group For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Preoperative Ketorolac For Participants With Renal Cell Carcinoma (RCC) | Control Group For Participants With Renal Cell Carcinoma (RCC)
Number analyzed (Participants) | 14 | 6 | 28 | 10
Participants | 0 | 0 | 2 | 2

2. Primary Outcome: Number of Participants Experiencing Clinically Significant Hematoma Development
Description: Post-surgical significant hematoma development is assessed as the number of participants experiencing a hematoma prior to hospital discharge.
Time Frame: Prior to Hospital Discharge (up to 13 days post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Ketorolac For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Control Group For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Preoperative Ketorolac For Participants With Renal Cell Carcinoma (RCC) | Control Group For Participants With Renal Cell Carcinoma (RCC)
Number analyzed (Participants) | 14 | 6 | 28 | 10
Participants | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants Returning to the Operating Room for Bleeding
Description: Post-operative bleeding is assessed at the number of participants needing to return to the operating room for bleeding, as determined by the treating surgeon.
Time Frame: Prior to Hospital Discharge (up to 13 days post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Ketorolac For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Control Group For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Preoperative Ketorolac For Participants With Renal Cell Carcinoma (RCC) | Control Group For Participants With Renal Cell Carcinoma (RCC)
Number analyzed (Participants) | 14 | 6 | 28 | 10
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Experiencing Postoperative Renal Failure
Description: Postoperative renal failure is assessed as the number of participants experiencing renal failure prior to hospital discharge.
Time Frame: Prior to Hospital Discharge (up to 13 days post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Ketorolac For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Control Group For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Preoperative Ketorolac For Participants With Renal Cell Carcinoma (RCC) | Control Group For Participants With Renal Cell Carcinoma (RCC)
Number analyzed (Participants) | 14 | 6 | 28 | 10
Participants | 0 | 0 | 0 | 1

5. Primary Outcome: Number of Participants Experiencing Postoperative Morbidity
Description: Postoperative morbidity is assessed as the count of participants experiencing at least one adverse event or serious adverse event from surgery to hospital discharge.
Time Frame: Prior to Hospital Discharge (up to 13 days post surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Ketorolac For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Control Group For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Preoperative Ketorolac For Participants With Renal Cell Carcinoma (RCC) | Control Group For Participants With Renal Cell Carcinoma (RCC)
Number analyzed (Participants) | 14 | 6 | 28 | 10
Participants | 6 | 1 | 14 | 6

6. Other Pre Specified Outcome: Transcriptome Analysis
Description: Transcriptome analysis will be performed to evaluate the effects of ketorolac on immune response pathways.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Flow Cytometry
Description: Flow Cytometry will be performed to evaluate the effects of ketorolac on immune response pathways.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

8. Other Pre Specified Outcome: T-Cell Receptor (TCR) Sequencing
Description: T-Cell receptor (TCR) sequencing will be performed to evaluate the effects of ketorolac on immune response pathways.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Single Cell RNA Sequencing
Description: Single cell RNA sequencing will be performed to evaluate the effects of ketorolac on immune response pathways.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Interleukin-1 Alpha (IL-1alpha) Levels
Description: IL-1alpha levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Interleukin-1beta (IL-1β) Levels
Description: IL-1beta levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Interleukin-2 (IL-2) Levels
Description: IL-2 levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Interleukin-6 (IL-6) Levels
Description: IL-6 levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Interleukin-8 (IL-8) Levels
Description: IL-8 levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Interleukin-10 (IL-10) Levels
Description: IL-10 levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Interleukin-12p70 (IL-12p70) Levels
Description: IL-12p70 levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Tumor Necrosis Factor-alpha (TNF-alpha) Levels
Description: TNF-alpha levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Interferon (INF)-Gamma Levels
Description: INF-gamma levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) Levels
Description: GM-CSF levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Monocyte Chemotactic and Activating Factor (MCAF) Levels
Description: MCAF levels will be compared between study arms.
Time Frame: Baseline, Day 1, Day 3 (if admitted to hospital), Day 7, Day 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information about adverse events was collected from the time of the preoperative visit through 28 days after surgery (up to 141 days), from participants who began study activities (had their standard of care surgery, and were administered ketorolac if they were randomized to the ketorolac study arm).
Arm/Group | Preoperative Ketorolac For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Control Group For Participants With Non-small Cell Lung Carcinoma (NSCLC) | Preoperative Ketorolac For Participants With Renal Cell Carcinoma (RCC) | Control Group For Participants With Renal Cell Carcinoma (RCC)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6 | 0/28 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/6 | 1/28 | 2/10
Other Adverse Events (participants affected / at risk) | 6/14 | 1/6 | 16/28 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative Ketorolac For Participants With Non-small Cell Lung Carcinoma (NSCLC) (N=14) | Control Group For Participants With Non-small Cell Lung Carcinoma (NSCLC) (N=6) | Preoperative Ketorolac For Participants With Renal Cell Carcinoma (RCC) (N=28) | Control Group For Participants With Renal Cell Carcinoma (RCC) (N=10)
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Hypotension (General disorders) | 0 | 0 | 1 | 0
Elevated cardiac troponin (Cardiac disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Subcutaneous emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative Ketorolac For Participants With Non-small Cell Lung Carcinoma (NSCLC) (N=14) | Control Group For Participants With Non-small Cell Lung Carcinoma (NSCLC) (N=6) | Preoperative Ketorolac For Participants With Renal Cell Carcinoma (RCC) (N=28) | Control Group For Participants With Renal Cell Carcinoma (RCC) (N=10)
Hematoma (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Thrombophlebitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Hypertension (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypotension (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Nausea/vomiting (Gastrointestinal disorders) | 1 | 0 | 10 | 6
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Belching/bloating (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Bowel obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dizziness (General disorders) | 0 | 0 | 1 | 0
Allergic reaction to oxycodone (General disorders) | 0 | 0 | 0 | 1
Edema (General disorders) | 0 | 0 | 1 | 1
Fever (General disorders) | 0 | 0 | 2 | 0
External ear pain (General disorders) | 0 | 0 | 1 | 0
Eye irritation (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Hyperglycemia (Endocrine disorders) | 0 | 0 | 1 | 0
Hyperglycemia (Endocrine disorders) | 0 | 0 | 0 | 1
Itching (General disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Tremor (General disorders) | 0 | 0 | 2 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Numbness (right hand) (General disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
High chest tube output (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Persistent air leak (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rib cage pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Low urine output (Renal and urinary disorders) | 0 | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT04495894/Prot_SAP_000.pdf